CLINICAL TRIAL: NCT00348296
Title: A Randomized, Double-blind, Placebo-controlled Multi-center Study of GB-0998 for Treatment of Systemic Sclerosis
Brief Title: Efficacy and Safety Study of GB-0998 for Treatment of Systemic Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Benesis Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0998-A1
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Last update posted 2010-07-30 (Estimated); Status verified 2010-07

CONDITIONS: Scleroderma, Systemic
Keywords: Scleroderma, Systemic
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Immunoglobulins, Intravenous

INTERVENTIONS:
Drug: High-dose intravenous immunoglobulin (Venoglobulin-IH)

SUMMARY:
This randomized, double-blind, placebo-controlled multi-center study will carry out to assess the efficacy of GB-0998 in the treatment of the systemic sclerosis based on the changes in modified Rodnan total skin thickness score (TSS) as primary endopoint, and in addition, to assess the safety of GB-0998.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have sclerosis located proximal to the elbow joint with diffused systemic scleroderma.
* Patients who have not less than 20 points of TSS.
* Patients with no appropriate therapeutic treatment.

Exclusion Criteria:

* Patients with severe hepatic disorder, severe renal disorder or severe heart disorder.
* Patients with malignant tumors.
* Patients who have the anamnesis of shock or hypersensitivity to this drug.
* Patients who have the anamnesis of cerebral infarction or symptom of these diseases.
* Patients who have been diagnosed as IgA deficiency in their past history.
* Pregnant, lactating, and probably pregnant patients, and patients who want to become pregnant.
* Patients who had any dose increase or new dosing of steroid within 12 weeks before consent.
* Patients who were administered other investigational drug within 12 weeks before consent.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Changes in TSS at 12 weeks

SECONDARY OUTCOMES:
Changes in joint motion, oral aperture, active hand spread, fingertip-to-palm distance, health assessment questionnaire, histological analysis of dermal section at 12 weeks.; Adverse events and laboratory test.

CONTACTS AND LOCATIONS:
Overall Officials: Kazuhiko Takehara, Professor, Study Chair — Kanazawa University
Locations (1):
- Nagasaki University, Nagasaki, Nagasaki, Japan

REFERENCES:
- [Derived] Takehara K, Ihn H, Sato S. A randomized, double-blind, placebo-controlled trial: intravenous immunoglobulin treatment in patients with diffuse cutaneous systemic sclerosis. Clin Exp Rheumatol. 2013 Mar-Apr;31(2 Suppl 76):151-6. Epub 2013 Jul 23. PMID 23910617